CLINICAL TRIAL: NCT05931822
Title: Quantitative Evaluation of Silver Diamine Fluoride Modified Restoration In Treating Hypomineralized First Permanent Molar In A Group Of Children"-A Clinical Study
Brief Title: Silver Diamine Fluoride Modified Restoration In Treating Hypomineralized First Permanent Molar.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Aya Ehab, Assistant lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A05031219
Record Dates: First submitted 2023-06-22; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Molar Incisor Hypomineralization
Keywords: MIH, silver diamine fluoride, children, glass ionomer
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver Diamine fluoride modified glass ionomer restoration (Active Comparator)
  Interventions: Other: Silver Diamine Fluoride 38%
- fluoride varnish and glass ionomer restoration (Active Comparator)
  Interventions: Other: fluoride varnish

INTERVENTIONS:
Other: Silver Diamine Fluoride 38% — silver diamine fluoride 38% brushed on the cavity for 1 minute before adding high viscosity glass ionomer restoration in one molar
  Arms: Silver Diamine fluoride modified glass ionomer restoration
Other: fluoride varnish — fluoride varnish brushed after adding the high viscosity glass ionomer restoration in the contralateral molar
  Arms: fluoride varnish and glass ionomer restoration

SUMMARY:
A randomized clinical trial to compare silver modified glass ionomer restorations to non silver glass ionomer restorations in hypo-mineralized first permanent molars in children and to measure the amount of wear of restoration in both groups along with detecting changes in hypersensitivity in hypomineralized molars in both groups after one year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral first permanent molars affected with molar incisor hypomineralization and with the same ICDAS II score.
* Both chosen molars should be of the same degree of MIH severity.

Exclusion Criteria:

* signs and symptoms of irreversible pulpitis or pulp necrosis.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Measuring surface wear using CAD-CAM software program | after 1 year
  impressions were taken after treatment and after one year the two impressions were scanned. The scans were superimposed to compare the surface change. T o standardize the measurements specific selected points on the occlusal surface was used.
Restoration Survival evaluation using the Atraumatic Restorative Treatment(ART) criteria | 1 year
  ART criterion was used to evaluate the restorations done after treatment then once again after one year.

SECONDARY OUTCOMES:
Tooth hypersensitivity was evaluated with Schiff cold air sensitivity scale (SCASS) | after 1 year
  The molars that were selected for treatment were tested for hypersensitivity. The air was delivered from a standard dental unit air syringe for 1 second at a distance of 1 cm and perpendicular to the occlusal surface of the tooth, before treatment ,after 1 week, 6 months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Abd Elatiif, professor, Study Director — Mansoura University, Mansoura, Egypt
Locations (1):
- Mansoura University, Al Mansurah, Dakaleya, Egypt

IPD SHARING:
Plan to Share IPD: No
my research is still under publishing and i am planning to get published within 1-2 months. Data in my research can be shared afterwards.

REFERENCES:
- [Derived] Saad AE, Alhosainy AY, Abdellatif AM. "Evaluation of Silver Diamine Fluoride Modified Atraumatic Restorative Treatment (SMART) on hypomineralized first permanent molar"- a randomized controlled clinical study. BMC Oral Health. 2024 Oct 4;24(1):1182. doi: 10.1186/s12903-024-04860-z. PMID 39367399